CLINICAL TRIAL: NCT03138980
Title: Mobile Self-Management of Irritable Bowel Syndrome for Adolescents: Pilot Study
Brief Title: Mobile Self-Management of Irritable Bowel Syndrome for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: BodiMojo, Inc. (Other)
Responsible Party: Principal Investigator, Lonnie Zeltzer, Professor, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-001825
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Irritable Bowel Syndrome; Abdominal Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile application (Experimental)
  Interventions: Behavioral: BodiMojo Buddy for IBS

INTERVENTIONS:
Behavioral: BodiMojo Buddy for IBS — Mobile application focusing on emotional coping skills for teens and young adults with IBS. Components of the module include: mood recorder and "mood cloud," with supportive feedback given based on mood choice; health behavior change support messages informed by mindfulness and self-compassion; quizzes with tailored feedback; library of meditations; an interactive coping skills advice section; and a link to an optional social support feature.

SUMMARY:
The objective of the proposed research is to conduct user testing of a mobile-based self-management support intervention for adolescents and young adults with Irritable Bowel Syndrome (IBS), a chronic digestive condition. The application (app; BodiMojo Buddy) uses a virtual coach that can serve to increase patient engagement through interactive skill-building, self-care, and mindfulness-based cognitive behavioral activities. If the BodiMojo Buddy mobile app is successful, it will have a significant public health impact by providing a mobile resource to the 10-15% of the US population who suffer from IBS and potentially improving health outcomes and reducing significant costs to the US healthcare system.

Study participation involves participants downloading and using the app for 30 days. During the 30 days, participants will interact with the app by inputting their current mood, receiving supportive feedback from the app, reading messages, and doing brief activities (such as relaxation activities, etc.). Before and after the 30 days of user testing, participants will complete a few brief questionnaires about their behavior, how their symptoms affect their life, and how they receive support from others. These questions will take around 20 minutes to complete at each administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-21 years
2. For adolescents: Parent-reported physician diagnosis of IBS, using pediatric Rome III diagnostic criteria for functional gastrointestinal disorders. For young adults: self-reported physician diagnosis of IBS using Rome III diagnostic criteria, or meeting criteria for IBS or functional abdominal pain as determined during phone screening.
3. Have daily use of an iPhone or iPad that meets the following technical specifications: at least iOS 8; for iPhones, must be iPhone 5 or above.
4. Able and willing to give informed assent/consent and comply with study requirements
5. Have one caregiver willing and able to participate in the study [only for 13-17 year olds]

Exclusion Criteria:

1. Inability to provide informed assent/permission/consent
2. Inability to read, speak, and understand English (because the app content/parent guides are written in English, as are the measures being used in the study)

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01-30 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-09-22 (Actual)

PRIMARY OUTCOMES:
Ratio of the days during the 30-day intervention period during which participants use the app | 30 days (from day 1 through day 30 of the 30-day intervention period)
  Determined by how often adolescents engaged and used certain features. To be considered feasible, teens must have opened the app on at least two-thirds of the days.
Acceptance | Within 7 days of competing the intervention
  Determined by participants' responses to acceptance test questions in the following domains: (1) perceived connectedness with the Buddy; (2) relevance of the self-management skill building content; and (3) usefulness of self-management skill-building content for IBS. Responses will be given on a one to seven-point-scale ranging "terrible" to "excellent." The intervention will be deemed acceptable if at least 80% of participants rate each question an average of at least "5" ("good") on the 7-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Pediatric Pain Program Research Offices, Los Angeles, California, United States